CLINICAL TRIAL: NCT07339787
Title: Diagnosis of Transient Ischemic Attacks in the Emergency Department
Acronym: DAITSU
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9766
Record Dates: First submitted 2026-01-05; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Transient Ischemic Attack; Cardiovascular Morbidity
Keywords: Transient Ischemic Attack; Cardiovascular Morbidity
MeSH Terms: conditions — Ischemic Attack, Transient

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients presenting a Transient Ischemic Attack (TIA) and admitted to the Emergency Department should be referred to a neurovascular specialist. In recent years, several hospitals have established TIA clinics. These units are day hospitals where all the necessary examinations are performed. Access to this expertise has proven beneficial in reducing cardiovascular morbidity and mortality, particularly the risk of early recurrence. Unfortunately, this access is limited by issues of medical demographics and unequal access to the healthcare system. In practice, this ideal care is not always possible. A portion of the TIA population is at low risk, and diagnostic and therapeutic interventions are limited, not always requiring neurovascular expertise.

The hypothesis of this research is that the management of a patient who has suffered a TIA (additional examinations, treatment, referral) is not linked to their cardiovascular risk and that the performance of additional examinations and therapies is incomplete.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years old)
* Having consulted the emergency department or been diagnosed with TIA during the period from January 1, 2024, to December 12, 2024 (records will be compiled via coding at the East Rescue regional emergency observatory)
* TIA will be defined as a sudden, transient neurological deficit that had disappeared by the time of arrival at the emergency department

Exclusion Criteria:

- Subjects with a suspected diagnosis of TIA, i.e., with a sudden, transient neurological deficit that had disappeared by the time of arrival at the emergency department.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (≥18 years old) having consulted the emergency department or been diagnosed with TIA during the period from January 1, 2024, to December 12, 2024 (records will be compiled via coding at the East Rescue regional emergency observatory)
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-02-06 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01-06 (Estimated)

PRIMARY OUTCOMES:
ABCD2 Score | Up to 12 months
  The ABCD2 score is a medical tool used by doctors after a TIA (Transient Ischemic Attack).
  The total score ranges from 0 to 7:
  * 0-3: low risk
  * 4-5: moderate risk
  * 6-7: high risk

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Urgences Médico-Chirurgicales Adules - CHU de Strasbourg - France, Strasbourg, France